CLINICAL TRIAL: NCT04936139
Title: Effectiveness of Art Therapy in the Level of Anxiety and Depression of Cancer Patients. Multicentric Random Clinical Trial (ATANDEC)
Brief Title: Art Therapy Effectiveness in the Level of Anxiety and Depression of Cancer Patients
Acronym: ATANDEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elisenda Campreciós Suñol (Other)
Collaborators: Fundació privada Nous Cims (Unknown); Althaia Xarxa Assistencial Universitària de Manresa (Other)
Responsible Party: Sponsor-Investigator, Elisenda Campreciós Suñol, Principal Investigator (Bachelor's in Nursing, MSc), Althaia Xarxa Assistencial Universitària de Manresa
Organization: Althaia Xarxa Assistencial Universitària de Manresa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEI 20/69
Record Dates: First submitted 2021-06-14; First posted 2021-06-23 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Cancer
Keywords: Art Therapy; Depression; Anxiety; Quality of Life; Coping Skills
MeSH Terms: conditions — Neoplasms; Depression; Anxiety Disorders | interventions — Art Therapy

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, parallel and multi-centric non-pharmacological clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Art Therapy (Experimental): Patients assigned to the intervention group will participate in 12 weekly group therapy workshop sessions.
  Interventions: Behavioral: Art Therapy
- Control group (No Intervention): Patients assigned to the control group will receive the usual follow-up care of each center provided for the cancer patient and will not perform art therapy workshops.
  They will be offered the opportunity to participate in the workshops once they have completed their participation in the study, putting them on a waiting list.

INTERVENTIONS:
Behavioral: Art Therapy — During the 12 planned sessions, different artistic disciplines will be used: visual arts, music, play, narrative, dramatization, movement and body expression.
  Each session is structured in 3 phases:
  i. A first part of encounter and contextualization, to make contact with oneself, with the art therapist and with the group through a relaxation or meditation activity (35 minutes).
  ii. A second part, where the session continues with the work of artistic elaboration and production with the different materials and the different artistic languages (50 minutes).
  iii. A third part where the participants will be invited to make a closing, a moment to welcome and share whoever wishes, the experiences that have been experienced. A dialogue is created between Work-Patient-Art Therapist (35 minutes).
  Arms: Art Therapy

SUMMARY:
Having a diagnosis of cancer leaves a great emotional impact when it comes to strategies for coping with illness and life after illness. Participation in an art therapy program to forge and improve the emotional well-being is considered.

Art therapy can be an effective intervention to help cancer patients lower their levels of anxiety and depression and in return improve their quality of life and their ability to cope with the disease.

DETAILED DESCRIPTION:
Introduction: The passage of a cancer through a person leaves a great emotional impact when it comes to strategies for coping with illness and life after illness. Participation in an art therapy program to forge and improve your emotional well-being is considered.

Research Project Hypothesis: Art therapy can be an effective intervention to help cancer patients lower their levels of anxiety and depression and in return improve their quality of life and their ability to cope with the disease.

Objectives: To evaluate the effectiveness of art therapy in reducing the levels of anxiety and depression in cancer patients, as well as in improving the quality of life and coping strategies.

Methodology: Randomized, controlled, parallel and multi-centric non-pharmacological clinical trial. Eight centers will participate in the study with an N of 423 patients. Patients older than 18 years of age who are diagnosed with cancer at any stage of treatment with the intention of radical treatment or palliative treatment with a life expectancy of more than 12 months will be included. If it is carried out in an online format, the person must have access to the internet. Patients who suffer from a current or previous serious psychological / psychiatric illness or those who have participated in an art therapy program structured in the context of oncological process will be excluded. Patients will be assigned to the control group (they will receive the usual follow-up from the center) or to the intervention group (art therapy program). Patients assigned to the intervention group will participate in an art therapy workshop once a week for 12 weeks, which will be done in person / online depending on the epidemiological situation of covid-19 and the needs of each center, The group will maintain the format (online / face-to-face) with which it has started throughout all the sessions.

Art therapy is a discipline that offers a space to meet with oneself, where one can dialogue with different artistic languages, with the aim of promoting emotional integration and looking for new ways to integrate difficult experiences through creative language.

Assessing anxiety and depression with the HAD scale, coping strategies with the Mini-MAC scale, and WHOQOL-BREF for quality of life will be used. Statistical analysis will be for treatment purposes. IBM SPSS Statistics v.24 and STATA v.14 will be used.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Intention for radical treatment or palliative treatment with a life expectancy of more than 12 months
* Have internet access in case the intervention is done online
* Agree to participate and sign informed consent

Exclusion Criteria:

* Patient with active diagnosis or personal history of severe psychological / psychiatric illness
* Patient who has participated in an art therapy program structured in the context of the oncological process

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2021-02-21 (Actual); Primary Completion 2023-11-03 (Actual); Study Completion 2023-11-03 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale (HAD scale) | 3 months
  The scale consists of 14 items that assess symptoms of anxiety and depression on a Likert scale of 4 response options. Scores between 0 and 7 are considered normal; between 8 and 10 doubtful, and scores above 11 for clinical problem of depression or anxiety.
Hospital Anxiety and Depression Scale (HAD scale) | 6 months
  The scale consists of 14 items that assess symptoms of anxiety and depression on a Likert scale of 4 response options. Scores between 0 and 7 are considered normal; between 8 and 10 doubtful, and scores above 11 for clinical problem of depression or anxiety.

SECONDARY OUTCOMES:
World Health Organization Quality of Life (WHOQOL-BREF scale) | 3 months
  The questionnaire contains a total of 26 questions, two global quality of life and general health questions, and one question from each of the 24 facets contained in the WHOQOL-100. It also consists of 4 areas or dimensions: physical health, psychological, social relationships and environment. Each item has 5 ordinary Likert-type response options and the time it takes is two weeks. Higher scores indicate better quality of life
World Health Organization Quality of Life (WHOQOL-BREF scale) | 6 months
  The questionnaire contains a total of 26 questions, two global quality of life and general health questions, and one question from each of the 24 facets contained in the WHOQOL-100. It also consists of 4 areas or dimensions: physical health, psychological, social relationships and environment. Each item has 5 ordinary Likert-type response options and the time it takes is two weeks. Higher scores indicate better quality of life
Mini-Mental Adjustment to Cancer Scale (MINI-MAC) | 3 months
  MINI-MAC is a 29-item instrument on a 4-choice Likert scale that assesses cognitive and behavioral responses to cancer. Differentiate 5 modes of coping: helplessness / hopelessness (ID), anxious worry (PA), cognitive avoidance (EN), fighting spirit (EL), and fatalism (FAE). Results are calculated for each of the examined strategies. Each strategy includes seven relevant statements. Every analysed subscale result range may be from 7 to 28. The higher the score, the stronger the behaviour typical for a given strategy of coping with càncer.
Mini-Mental Adjustment to Cancer Scale (MINI-MAC) | 6 months
  MINI-MAC is a 29-item instrument on a 4-choice Likert scale that assesses cognitive and behavioral responses to cancer. Differentiate 5 modes of coping: helplessness / hopelessness (ID), anxious worry (PA), cognitive avoidance (EN), fighting spirit (EL), and fatalism (FAE). Results are calculated for each of the examined strategies. Each strategy includes seven relevant statements. Every analysed subscale result range may be from 7 to 28. The higher the score, the stronger the behaviour typical for a given strategy of coping with càncer.

CONTACTS AND LOCATIONS:
Overall Officials: Pau Gomes, MsC, Study Chair — Fundació Nou Cims
Locations (1):
- Althaia Xarxa Assistencial Universitària de Manresa, Manresa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Archer S, Buxton S, Sheffield D. The effect of creative psychological interventions on psychological outcomes for adult cancer patients: a systematic review of randomised controlled trials. Psychooncology. 2015 Jan;24(1):1-10. doi: 10.1002/pon.3607. Epub 2014 Jun 21. PMID 24953449
- [Result] Andreu Vaillo Y, Murgui Perez S, Martinez Lopez P, Romero Retes R. Mini-Mental Adjustment to Cancer Scale: Construct validation in Spanish breast cancer patients. J Psychosom Res. 2018 Nov;114:38-44. doi: 10.1016/j.jpsychores.2018.09.004. Epub 2018 Sep 15. PMID 30314577
- [Result] Oster I, Svensk AC, Magnusson E, Thyme KE, Sjodin M, Astrom S, Lindh J. Art therapy improves coping resources: a randomized, controlled study among women with breast cancer. Palliat Support Care. 2006 Mar;4(1):57-64. doi: 10.1017/s147895150606007x. PMID 16889324
- [Result] Krikorian A, Limonero JT, Mate J. Suffering and distress at the end-of-life. Psychooncology. 2012 Aug;21(8):799-808. doi: 10.1002/pon.2087. Epub 2011 Oct 11. PMID 21990213
- [Result] Monti DA, Peterson C, Kunkel EJ, Hauck WW, Pequignot E, Rhodes L, Brainard GC. A randomized, controlled trial of mindfulness-based art therapy (MBAT) for women with cancer. Psychooncology. 2006 May;15(5):363-73. doi: 10.1002/pon.988. PMID 16288447
- [Result] Puetz TW, Morley CA, Herring MP. Effects of creative arts therapies on psychological symptoms and quality of life in patients with cancer. JAMA Intern Med. 2013 Jun 10;173(11):960-9. doi: 10.1001/jamainternmed.2013.836. PMID 23699646
- [Result] Svensk AC, Oster I, Thyme KE, Magnusson E, Sjodin M, Eisemann M, Astrom S, Lindh J. Art therapy improves experienced quality of life among women undergoing treatment for breast cancer: a randomized controlled study. Eur J Cancer Care (Engl). 2009 Jan;18(1):69-77. doi: 10.1111/j.1365-2354.2008.00952.x. PMID 19473224
- [Result] Thyme KE, Sundin EC, Wiberg B, Oster I, Astrom S, Lindh J. Individual brief art therapy can be helpful for women with breast cancer: a randomized controlled clinical study. Palliat Support Care. 2009 Mar;7(1):87-95. doi: 10.1017/S147895150900011X. PMID 19619378
- [Result] Xu L, Cheng P, Wu Y, Zhang J, Zhu J, Cui J, Yu R. The effects of art therapy on anxiety and depression in breast cancer patients: An updated meta-analysis. Eur J Cancer Care (Engl). 2020 Sep;29(5):e13266. doi: 10.1111/ecc.13266. Epub 2020 May 25. PMID 32452121
- [Result] Zhang MF, Wen YS, Liu WY, Peng LF, Wu XD, Liu QW. Effectiveness of Mindfulness-based Therapy for Reducing Anxiety and Depression in Patients With Cancer: A Meta-analysis. Medicine (Baltimore). 2015 Nov;94(45):e0897-0. doi: 10.1097/MD.0000000000000897. PMID 26559246
- [Result] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820